CLINICAL TRIAL: NCT00334971
Title: Aromatase Activity and Ovarian Growth Factors in Preovulatory Follicles
Brief Title: Aromatase Activity and Ovarian Growth Factors in African-American Versus Caucasian Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Janet E. Hall, MD, Associate Physician, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2002-P-001354; Sundry (Other: MGH-REU)
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Healthy; Fragile X Syndrome
Keywords: African-American; estradiol; luteinizing hormone; follicle stimulating hormone; androstenedione; aromatase; inhibins; ovarian; Healthy volunteers; Fragile X
MeSH Terms: conditions — Fragile X Syndrome | interventions — Oocyte Retrieval

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Other): Healthy Caucasian women 18-35 years old
  Interventions: Procedure: Follicle Aspiration
- 2 (Other): Healthy African-American women 18-35 years old
  Interventions: Procedure: Follicle Aspiration
- 3 (Other): Healthy Caucasian women 36-45 years old
  Interventions: Procedure: Follicle Aspiration
- 4 (Other): Female fragile X premutation carriers 18-45 years old
  Interventions: Procedure: Follicle Aspiration

INTERVENTIONS:
Procedure: Follicle Aspiration — Follicles will be aspirated using a transvaginal ultrasound guided needle.

SUMMARY:
The purpose of the study is to understand how the ovarian follicle (the fluid filled structure in the ovary that contains the egg) makes estrogen and other hormones during normal aging, in women with different ethnic backgrounds, and in Fragile X premutation carriers.

During reproductive aging, estradiol levels are increased, a phenomenon that may be related to increased aromatase activity. The investigators' own preliminary data suggest that estradiol is increased in African-American women compared to Caucasian women, which may also be related to aromatase activity. In addition, the investigators have examined female fragile X premutation carriers who still have regular menstrual cycles and have demonstrated evidence of early ovarian aging compared to age-matched controls.

**WE ARE RECRUITING ONLY WOMEN WITH FRAGILE-X PREMUTATION**

DETAILED DESCRIPTION:
The purpose of the study is to examine intrafollicular changes in aromatase and ovarian growth factors in reproductive aged women,African-American women compared to Caucasian controls, and Fragile X premutation carriers.

Hypotheses:

* Aromatase activity is up-regulated in preovulatory follicles with aging, accounting for the increased estradiol levels in the face of decreased inhibin secretion in reproductive aging.
* Increased estradiol in the face of normal inhibin A and inhibin B suggests up-regulation of aromatase in African-American women.
* Aromatase activity is down-regulated in preovulatory follicles in fragile X premutation carriers compared to age-matched controls and the activity is associated with FMR1 mRNA levels.

ELIGIBILITY:
Inclusion Criteria:

Reproductively Younger Non-African-American Women:

* 18-35 years of age
* Body mass index (BMI) less than or equal to 30
* Regular menstrual cycles (25-35 days long)
* Negative beta-human chorionic gonadotrophin (HCG)
* Normal prolactin and thyroid stimulating hormone (TSH) levels
* Hemoglobin greater than or equal to 11.0 gm/dl
* Luteal phase progesterone level indicating ovulation on a previous cycle (> 3 ng/ml)
* Not currently trying to get pregnant
* No blood donations within 2 months of initiating the blood sampling portion of the study
* On no medications thought to interfere with normal menstrual cycle dynamics
* Not current smokers or no exposure to passive smoke in the home or workplace (greater than 8 hours per day with a smoker of > 10 cigarettes per day)
* Normal platelet count and PT/PTT
* No history of pelvic adhesions and accessible ovarian position as assessed by transvaginal ultrasound

Reproductively Younger African-American Women:

* 18-35 years of age
* Meets all other inclusion criteria for the reproductively younger non-African-American population outlined above

Reproductively Older Non-African-American Women:

* 36-45 years of age
* Meets all other inclusion criteria for the reproductively younger non-African-American population outlined above.

Reproductive Aged Fragile X Premutation Carriers

* Fragile X premutation carriers, with FMR1 CGG repeat lengths between 41 and 200.
* 18-45 years of age
* Meets all other inclusion criteria for the reproductively younger non-African-American population outlined above.

Exclusion Criteria:

* Hemoglobin level less than 11 gm/dl at time of screening

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2004-09; Primary Completion 2012-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Serum androstenedione, E2, A/E2, inhibin A, and inhibin B | at first day of menses until day after aspiration procedure
Follicular fluid androstenedione, E2, A/E2, inhibin A, and inhibin B | after aspiration procedure
RT-PCR results for aromatase in aspirated follicular fluid, when follicle is > 14 mm | after aspiration procedure

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Hall, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Reproductive Endocrine Unit, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Welt CK, McNicholl DJ, Taylor AE, Hall JE. Female reproductive aging is marked by decreased secretion of dimeric inhibin. J Clin Endocrinol Metab. 1999 Jan;84(1):105-11. doi: 10.1210/jcem.84.1.5381. PMID 9920069
- [Background] Santoro N, Brown JR, Adel T, Skurnick JH. Characterization of reproductive hormonal dynamics in the perimenopause. J Clin Endocrinol Metab. 1996 Apr;81(4):1495-501. doi: 10.1210/jcem.81.4.8636357.
- [Background] Reame NE, Kelche RP, Beitins IZ, Yu MY, Zawacki CM, Padmanabhan V. Age effects of follicle-stimulating hormone and pulsatile luteinizing hormone secretion across the menstrual cycle of premenopausal women. J Clin Endocrinol Metab. 1996 Apr;81(4):1512-8. doi: 10.1210/jcem.81.4.8636360.
- [Background] Klein NA, Battaglia DE, Fujimoto VY, Davis GS, Bremner WJ, Soules MR. Reproductive aging: accelerated ovarian follicular development associated with a monotropic follicle-stimulating hormone rise in normal older women. J Clin Endocrinol Metab. 1996 Mar;81(3):1038-45. doi: 10.1210/jcem.81.3.8772573.
- [Background] MacNaughton J, Banah M, McCloud P, Hee J, Burger H. Age related changes in follicle stimulating hormone, luteinizing hormone, oestradiol and immunoreactive inhibin in women of reproductive age. Clin Endocrinol (Oxf). 1992 Apr;36(4):339-45. doi: 10.1111/j.1365-2265.1992.tb01457.x. PMID 1424166
- [Background] Burger HG, Dudley EC, Hopper JL, Shelley JM, Green A, Smith A, Dennerstein L, Morse C. The endocrinology of the menopausal transition: a cross-sectional study of a population-based sample. J Clin Endocrinol Metab. 1995 Dec;80(12):3537-45. doi: 10.1210/jcem.80.12.8530596.
- [Background] Welt CK, Smith ZA, Pauler DK, Hall JE. Differential regulation of inhibin A and inhibin B by luteinizing hormone, follicle-stimulating hormone, and stage of follicle development. J Clin Endocrinol Metab. 2001 Jun;86(6):2531-7. doi: 10.1210/jcem.86.6.7597. PMID 11397851
- [Background] Schneyer AL, Fujiwara T, Fox J, Welt CK, Adams J, Messerlian GM, Taylor AE. Dynamic changes in the intrafollicular inhibin/activin/follistatin axis during human follicular development: relationship to circulating hormone concentrations. J Clin Endocrinol Metab. 2000 Sep;85(9):3319-30. doi: 10.1210/jcem.85.9.6767. PMID 10999828
- [Background] Khoury MJ, Erickson JD. Maternal factors in dizygotic twinning: evidence from interracial crosses. Ann Hum Biol. 1983 Sep-Oct;10(5):409-15. doi: 10.1080/03014468300006601. PMID 6638936
- [Background] KNOX G, MORLEY D. Twinning in Yoruba women. J Obstet Gynaecol Br Emp. 1960 Dec;67:981-4. doi: 10.1111/j.1471-0528.1960.tb09255.x. No abstract available. PMID 13757217
- [Background] Myrianthopoulos NC. An epidemiologic survey of twins in a large, prospectively studied population. Am J Hum Genet. 1970 Nov;22(6):611-29. No abstract available. PMID 5518457
- [Background] Martin NG, Robertson DM, Chenevix-Trench G, de Kretser DM, Osborne J, Burger HG. Elevation of follicular phase inhibin and luteinizing hormone levels in mothers of dizygotic twins suggests nonovarian control of human multiple ovulation. Fertil Steril. 1991 Sep;56(3):469-74. doi: 10.1016/s0015-0282(16)54542-7. PMID 1894024
- [Background] Faerstein E, Szklo M, Rosenshein NB. Risk factors for uterine leiomyoma: a practice-based case-control study. II. Atherogenic risk factors and potential sources of uterine irritation. Am J Epidemiol. 2001 Jan 1;153(1):11-9. doi: 10.1093/aje/153.1.11. PMID 11159140
- [Background] Sondik EJ. Breast cancer trends. Incidence, mortality, and survival. Cancer. 1994 Aug 1;74(3 Suppl):995-9. doi: 10.1002/1097-0142(19940801)74:3+3.0.co;2-m. PMID 8039156
- [Background] Perry HM 3rd, Horowitz M, Morley JE, Fleming S, Jensen J, Caccione P, Miller DK, Kaiser FE, Sundarum M. Aging and bone metabolism in African American and Caucasian women. J Clin Endocrinol Metab. 1996 Mar;81(3):1108-17. doi: 10.1210/jcem.81.3.8772584.
- [Background] Woods MN, Barnett JB, Spiegelman D, Trail N, Hertzmark E, Longcope C, Gorbach SL. Hormone levels during dietary changes in premenopausal African-American women. J Natl Cancer Inst. 1996 Oct 2;88(19):1369-74. doi: 10.1093/jnci/88.19.1369. PMID 8827014
- [Background] Woods MN, Gorbach SL, Longcope C, Goldin BR, Dwyer JT, Morrill-LaBrode A. Low-fat, high-fiber diet and serum estrone sulfate in premenopausal women. Am J Clin Nutr. 1989 Jun;49(6):1179-83. doi: 10.1093/ajcn/49.6.1179. PMID 2543203
- [Background] Manson JM, Sammel MD, Freeman EW, Grisso JA. Racial differences in sex hormone levels in women approaching the transition to menopause. Fertil Steril. 2001 Feb;75(2):297-304. doi: 10.1016/s0015-0282(00)01723-4. PMID 11172830
- [Background] Welt CK, Schneyer AL. Differential regulation of inhibin B and inhibin a by follicle-stimulating hormone and local growth factors in human granulosa cells from small antral follicles. J Clin Endocrinol Metab. 2001 Jan;86(1):330-6. doi: 10.1210/jcem.86.1.7107. PMID 11232020
- [Background] Welt CK, Lambert-Messerlian G, Zheng W, Crowley WF Jr, Schneyer AL. Presence of activin, inhibin, and follistatin in epithelial ovarian carcinoma. J Clin Endocrinol Metab. 1997 Nov;82(11):3720-7. doi: 10.1210/jcem.82.11.4345. PMID 9360531
- [Derived] Shaw ND, Srouji SS, Welt CK, Cox KH, Fox JH, Adams JM, Sluss PM, Hall JE. Evidence that increased ovarian aromatase activity and expression account for higher estradiol levels in African American compared with Caucasian women. J Clin Endocrinol Metab. 2014 Apr;99(4):1384-92. doi: 10.1210/jc.2013-2398. Epub 2013 Nov 27. PMID 24285681